CLINICAL TRIAL: NCT00547963
Title: Reducing Injury, ETOH and THC Use Among ED Patients
Brief Title: Brief Counseling to Reduce Injuries Among Emergency Department Patients Who Report Alcohol and Substance Use
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Janette Baird, PhD, Injury Prevention Center, Rhode Island Hospital, Brown University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA-BAI-013709; NIH Grant number 5R01AA013709
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Alcohol Drinking; Marijuana Smoking
Keywords: Alcohol Drinking; Marijuana Smoking; Substance Use; Emergency Department (ED)
MeSH Terms: conditions — Alcohol Drinking; Marijuana Smoking; Substance-Related Disorders; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): two brief counseling sessions delivered to ED patients who report conjoint alcohol and marijuana use
  Interventions: Behavioral: brief counseling

INTERVENTIONS:
Behavioral: brief counseling — baseline assessment + two 40 minute sessions of brief counseling

SUMMARY:
The purpose of this study is to determine the effectiveness of two brief counseling sessions delivered to emergency department (ED) patients who report conjoint alcohol and marijuana use, in reducing injuries and other negative consequences, in comparison to an assessment only group.

DETAILED DESCRIPTION:
Alcohol and substance use remain a significant predictor of injuries, health and psychosocial consequences.

ED patients who were not being treated for critical conditions were asked about their use of alcohol and marijuana. Patients who self-reported the use of both substances were asked to participate in the study.

Recruited participants were given a baseline assessment and then randomized a treatment or a control condition. The treatment condition consisted of two 40 minute sessions of brief counseling. The first session took place in the ED the second session occurred within two weeks of being seen in the ED.

Participants completed assessments three and twelve months after being recruited in the ED. The primary dependent variables for this study are 12 month injuries and self-reported levels of negative life consequences associated with alcohol and marijuana use.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18 years of age or older.
* Participants will have a current DSM-IV diagnosis of alcohol dependence.
* Participants will have signed a witnessed informed consent.

Exclusion Criteria:

* Participants who meet current DSM-IV criteria for bipolar disorder, schizophrenia, dementia, or a psychological disorder requiring medication.
* Participants who have had more than seven days of inpatient treatment for substance use disorders in the 30 days previous to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2003-12; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Substance use; injuries, alcohol and marijuana negative consequences | 3 and 12 months

SECONDARY OUTCOMES:
Mediators and moderators of treatment efficacy | 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Janette Baird, PhD, Principal Investigator — Injury Prevention Center, Rhode Island Hospital, Brown University
Locations (1):
- Injury Prevention Center, Rhode Island Hospital, Brown University, Providence, Rhode Island, United States